CLINICAL TRIAL: NCT05115149
Title: The Study on the еffectiveness of the Integration of a Device Based on a Neural Interface and Neurostimulation of the Spinal Cord in the Rehabilitation of Patients With Upper Limb Movement Impairments Due to Neurological Disorders.
Brief Title: The Study of a Neural Interface and a Neurostimulation in the Rehabilitation of Upper Limb Movement Impairments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Samara State Medical University (Other); Samara Regional Clinical Hospital V.D. Seredavin (Other); Kazan Federal University (Other); Far Eastern Federal University (Other); EirMED Rehabilitation Center (Unknown); Pavlov Institute of Physiology, Russian Academy of Science (Unknown); IT Universe LLC (Unknown); VIBRAINT RUS LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Skoltech-CNBR1
Record Dates: First submitted 2021-10-11; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Spinal Cord Injuries
Keywords: Stroke; Transcutaneous spinal cord stimulation; tSCS; Brain-computer interface; BCI; Spinal Cord Injuries; Rehabilitation
MeSH Terms: conditions — Stroke; Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are categorised by the type of injury (spinal cord injury or stroke) and by the rehabilitation stage (early stage, later stage). Within those categories participants are randomly assigned to experimental and delay (control) groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients rehabilitation outcomes will be assessed by blinded assessors. In Neva Arm some patients will receive sham tSCS, with gradient decrease of the stimulation intensity from threshold level to 0 during one minute, as described in PMID 29335430 and PMID: 31996455
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volga: tSCS during the exercise (Experimental): Stimulation during the excercise
  Interventions: Device: VIBRAINT RehUp robotic orthosis; Procedure: tSCS during the exercise; Device: Neostim-5; Procedure: Exercise
- Neva: tSCS prior to the exercise (Experimental): Stimulation prior to the action
  Interventions: Device: VIBRAINT RehUp robotic orthosis; Procedure: tSCS prior to the exercise; Device: Neostim-5; Procedure: Exercise

INTERVENTIONS:
Device: VIBRAINT RehUp robotic orthosis — VIBRAINT RehUp robotic orthosis is a robotic arm that supports movement of a paralyzed arm. The robotic device is connected to a BCI. VIBRAINT RehUp software decodes imagery of a movement of the paralyzed arm and/or selective attention to the target of movement.
Procedure: tSCS during the exercise — During the exercise transcutaneous stimulation of the spinal cord and, in some cases, peripheral nerves is also performed.
  tSCS is performed with the localization of electrodes between the spinous processes of the vertebrae C2-C3 and C5-C6, anodes - above the clavicles or above the crests of the iliac bones, bipolar or monopolar pulses with a frequency of 30 Hz, modulated with a frequency of 5 Hz.
  Arms: Volga: tSCS during the exercise
Procedure: tSCS prior to the exercise — Prior to the exercise transcutaneous stimulation of the spinal cord and, in some cases, peripheral nerves is also performed.
  tSCS is performed with the localization of electrodes between the spinous processes of the vertebrae C2-C3 and C5-C6, anodes - above the clavicles or above the crests of the iliac bones, bipolar or monopolar pulses with a frequency of 30 Hz, modulated with a frequency of 5 Hz.
  Arms: Neva: tSCS prior to the exercise
Device: Neostim-5 — Neostim-5 is intended for the transcutaneous spinal cord noninvasive stimulation from 0 up to 250 2 mA (step 1mA). Neostim allows to stimulate up to five different segments of spinal cord. The device can be synchronised with other devices.
Procedure: Exercise — The partcipant recieves a mental task - to imagine a movement or to concentrate on the goal. Upon successful completion of the given mental task, the VIBRAINT RehUp robotic exerciser moves the paralyzed limb. In the presence of muscular activity in a limb, an additional condition for the start of movement can be EMG activity in an agonist muscle assisting the robot movement.

SUMMARY:
The aim of the study is to investigate the effectiveness of a new rehabilitation technology for paralysis that occurs after stroke or spinal cord injury. The research will jointly use a prototype neurorehabilitation orthosis, in which a robotic device moves a paralyzed arm at the command of a non-invasive brain-computer interface to perform a game life-like task augmented using a virtual-reality display, as well as an electrical stimulation device that activates the spinal cord and/or muscles of the paralyzed arm.

Investigators expect that a portion of the patients participating in the study will have an improvement in arm mobility by the end of the study.

Participants who express their special written consent will have venous blood tests conducted three times for subsequent analysis of lipid biomarkers, in order to further evaluate the effectiveness of rehabilitation methods based on biochemical analysis.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effectiveness of a new rehabilitation technology for paralysis that occurs after stroke or spinal cord injury. The research will jointly use a prototype neurorehabilitation orthosis, in which a robotic device moves a paralyzed arm at the command of a non-invasive brain-computer interface to perform a game life-like task in virtual reality (for example, aiming a hand-held virtual toy gun at a target), as well as an electrical stimulation device that activates the spinal cord and/or muscles of the paralyzed arm.

The study is carried out to collect data on the role of central and spinal mechanisms in the plasticity of neuronal circuits that determine the effect of combined spinal neurostimulation and robotic rehabilitation under the control of non-invasive neural interfaces in patients in early and late rehabilitation period after acute cerebrovascular accident and in patients after trauma of the cervical and upper thoracic spinal cord.

The study will use two technologies - neural interfaces and transcutaneous electrical stimulation of the spinal cord. Neural interfaces are a rapidly developing area at the intersection of medicine, neuroscience, biology, engineering, robotics, physics, mathematics, and materials science, which aims to reproduce and supplement brain functions and correct these functions in cases of neurological lesions. The possibility of using neural interfaces for the treatment of neurological disorders, including disorders resulting from spinal cord and brain injuries, epilepsy, strokes, and neurodegenerative diseases, such as Parkinson's disease, has been demonstrated.

Transcutaneous spinal cord stimulation (tSCS) is a method for non-invasive control of the activity of human spinal neural networks used to restore locomotor functions after spinal cord injury (SCI). The published research results show that tSCS modulates the activity of not only spinal but also cortical neuronal networks.

It is expected that the use of tSCS in conjunction with the use of neural interfaces will increase the effectiveness of neural interfaces for the rehabilitation of neurological lesions, including stroke, and SCI.

Biochemical monitoring will be applied for objective monitoring of the physiological conditions of patients, such as the physiological state of muscle tissue and the level of neuropathic pain. This method is based on the identification of metabolic and lipid compounds associated with physiological parameters in blood plasma samples, and the subsequent use of these compounds as biomarkers to assess the effectiveness of rehabilitation techniques carried out using the neural interface, as well as to optimize them. This monitoring will be helpful for each individual patient, as it will provide additional information about the course of rehabilitation. Blood sampling and follow-up testing will only be performed for patients who gave their written consent for this procedure. The analysis results will be stored in anonymized form.

The study participants will receive up to 12 rehabilitation procedures, each lasting about one hour, within two-four weeks. During the procedure, the activity of the brain (electroencephalogram) and muscles (electromyogram) will be recorded using non- invasive electrodes placed on the scalp and body. Also, during the study, electrical stimulation will be performed with non-invasive electrodes placed on the body.

During the exercise, participants focus their attention on the target of movement and/or imagine that their arms perform a movement. If the task is completed correctly, the robot will move the arm towards the target. This movement can additionally be accompanied with functional electrical stimulation using disposable electrodes glued to the skin on the back and/or the arms. The strength of the stimulation will be adjusted so as not to cause discomfort. Participants will be randomly assigned to groups, and participants in some groups will receive tSCS and some will not.

On the day of inclusion in the study, as part of Visit 1 (screening), anamnesis will be collected, and there will be performed assessment on the study scales, BCI testing, an EMG study with registration of muscle activity (rhomboid, pectoralis major, biceps, deltoid) and / or visual determination of tSCS thresholds.

After Visit 1, patients in the study groups will undergo 12 procedures of BCI-driven robotic rehabilitation accompanied by tSCS.

Visit 2 is carried out the next day after the end of the study to assess the study scales and conduct the EMG study described above.

Visit 3 is carried out one month after the end of the study to assess the study scales and conduct an EMG study.

Throughout the study, adverse events (AEs) will be monitored. Sessions will be held daily in 6/1 or 5/2 mode, in a rehabilitation room or at patients' homes, with a session duration of about 60 minutes. The duration of Visits 1-3 will be approximately 2 hours.

Investigators expect that a portion of the patients participating in the study will have an improvement in voluntary arm movements by the end of the study.

Patient data will be recorded and stored in anonymized form. Only research team members will have access to this information. If it is necessary to publish individual results on study scales, diagnoses, anamnesis, and age of participants, participants will be identified with codes. The study data is supposed to be stored for 10 years on a protected file storage with limited access.

ELIGIBILITY:
Criteria for inclusion in the study of patients:

1. Signed written informed consent.
2. Men or women aged 18 to 60 years after a first occurred acute cerebrovascular accident or in the recovery period after injury of the cervical and upper thoracic spinal cord.
3. Early or late rehabilitation period of acute cerebrovascular accident by the type of ischemic stroke or the consequences of SCI in the late recovery period
4. Diagnosis of "acute ischemic cerebrovascular accident", or a condition after spinal cord injury at the C3-C7 level, moderate or high severity ASIA A and ASIA B, according to the discharge summary, MRI or CT.
5. For groups of patients with stroke: the degree of severity of paresis of the upper limb from 3 points to 0 (according to the 6-point MRC muscle strength scale https://cpd-program.ru/methods/mrc.htm)
6. The patient's ability and willingness to comply with the requirements of this protocol.
7. Expressed patient motivation for rehabilitation.

Inclusion criteria for healthy volunteers:

1. Signed written informed consent.
2. Men or women between the ages of 18 and 40
3. Absence of somatic and psychiatric diseases (according to the reports of the subject and according to the examination of a medical specialist before the start of the study)
4. Ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. Severe cognitive impairment (<10 points on the Montreal Cognitive Assessment Scale).
2. The score on the Hamilton scale is above 18 points.
3. The rating on the Rankin scale is higher than 4 points.
4. Concomitant diseases that cause a decrease in muscle strength or an increase in muscle tone in the upper limbs (for example, cerebral palsy, brain damage as a result of trauma) or rigidity (for example, Parkinson's disease, contracture).
5. Late stages of arthritis or significant limitation of range of motion.
6. The absence of a part of the upper limb due to amputation caused by various reasons.
7. Any medical condition, including mental illness or epilepsy, that may affect the interpretation of the test results, the conduct of the test, or the safety of the patient.
8. Alcohol abuse, medical marijuana use, or light drug use in the previous 12 months.
9. Use of experimental drugs or medical devices within the previous 30 days prior to Visit 1.
10. Inability to comply with research procedures, according to the researcher.
11. The severity of the patient's condition according to the data of the neurological or somatic status, which does not allow full rehabilitation
12. Visual acuity less than 0.2 in the weakest eye according to the table of visual acuity of Sivtsev.
13. Unstable angina and / or heart attack during the previous month
14. History of stroke (for patients with spinal cord injury) or recurrent stroke (for patients with acute cerebrovascular accident).
15. Uncontrolled arterial hypertension.
16. Ataxia.
17. Pacemaker and / or other implanted electronic devices.
18. Taking muscle relaxants.
19. Peripheral neuropathy.
20. Concomitant diseases in the stage of exacerbation or decompensation, requiring active therapy.
21. The presence of allergic reactions and / or other skin lesions at the place of application of the heart rate electrodes at the time of the study.
22. Acute urinary tract infections.
23. Acute thrombophlebitis.
24. All forms of epilepsy.
25. Benign and malignant neoplasms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer scale for the upper limb after the rehabilitation procedures | 2 weeks
  Dynamics according to the Fugl-Meyer Assessment for Upper Extremity parts A-D (FMA-UE A-D) that assesses motor function in a range from 0 (worst score) to 66 (best score). Details aviable at https://www.gu.se/en/neuroscience-physiology/fugl-meyer-assessment.
Change from Baseline Fugl-Meyer scale for the upper limb in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Fugl-Meyer Assessment for Upper Extremity parts A-D (FMA-UE A-D) that assesses motor function in a range from 0 (worst score) to 66 (best score). Details aviable at https://www.gu.se/en/neuroscience-physiology/fugl-meyer-assessment.
Change from Baseline Action Research Arm Test after the rehabilitation procedures | 2 weeks
  Dynamics according to the Action Research Arm Test (ARAT) that assesses motor function in a range from 0 (worst score) to 57 (best score). Details available at https://www.physiopedia.com/Action_Research_Arm_Test_(ARAT) .
Change from Baseline Action Research Arm Test in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Action Research Arm Test (ARAT) that assesses motor function in a range from 0 (worst score) to 57 (best score). Details available at https://www.physiopedia.com/Action_Research_Arm_Test_(ARAT) .

SECONDARY OUTCOMES:
Change from Baseline Accuracy of BCI tasks after the rehabilitation procedures | 2 weeks
  Dynamics of accuracy for BCI tasks (% of correctly completed tasks)
Change from Baseline in the Accuracy of BCI tasks in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics of accuracy for BCI tasks (% of correctly completed tasks)
Change from Baseline Rivermead Mobility Index after the rehabilitation procedures | 2 weeks
  Dynamics according to the Rivermead Mobility Index (RMI) that assesses overall mobility in a range from 0 (worst score) to 15 (best score). Details available at https://www.physio-pedia.com/Rivermead_Mobility_Index .
Change from Baseline Rivermead Mobility Index results in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Rivermead Mobility Index (RMI) that assesses overall mobility in a range from 0 (worst score) to 15 (best score). Details available at https://www.physio-pedia.com/Rivermead_Mobility_Index .
Change from Baseline Ashworth Spasticity Scale after the rehabilitation procedures | 2 weeks
  Dynamics according to the Ashworth Spasticity Scale that assesses spasticity in a range from 0 (best score) to 4 (worst score). Details available at https://www.sralab.org/rehabilitation-measures/ashworth-scale- modified-ashworth-scale .https://www.sralab.org/rehabilitation-measures/ashworth-scale- modified-ashworth-scale
Change from Baseline Ashworth Spasticity Scale in two four after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Ashworth Spasticity Scale that assesses spasticity in a range from 0 (best score) to 4 (worst score). Details available at https://www.sralab.org/rehabilitation-measures/ashworth-scale- modified-ashworth-scale.
Change from Baseline The Capabilities of Upper Extremity Test after the rehabilitation procedures | 2 weeks
  Dynamics according to the Capabilities of the Upper Extremity Test (CUE-T). CUE-T is a performance measure intended to assess upper extremity function following spinal cord injury. Minimum is 0 (worst score), maximum unilateral (arm + hand) converted score is 60 (best for one hand). Derails available at https://www.jefferson.edu/university/rehabilitation-sciences/departments/outcomes-measurement/measures-assessments/capabilities-of-the-upper-extremity-test-cue-t.html
Change from Baseline The Capabilities of Upper Extremity Test in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Capabilities of the Upper Extremity Test (CUE-T). CUE-T is a performance measure intended to assess upper extremity function following spinal cord injury. Minimum is 0 (worst score), maximum unilateral (arm + hand) converted score is 60 (best for one hand). Derails available at https://www.jefferson.edu/university/rehabilitation-sciences/departments/outcomes-measurement/measures-assessments/capabilities-of-the-upper-extremity-test-cue-t.html
Change from Baseline Spinal Cord Independence Measure III after the rehabilitation procedures | 2 weeks
  Dynamics according to the Spinal Cord Independence Measure III (SCIM III) that assesses a spinal cord injured patient's independence in a range from 0 (worst score) to 100 (best score). Details available at https://scireproject.com/wp- content/uploads/SCIM_Toolkit_Printable-1.pdf
Change from Baseline Spinal Cord Independence Measure III in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the Spinal Cord Independence Measure III (SCIM III) that assesses a spinal cord injured patient's independence in a range from 0 (worst score) to 100 (best score). Details available at https://scireproject.com/wp- content/uploads/SCIM_Toolkit_Printable-1.pdf
Change from Baseline NIH Stroke Scale after the rehabilitation procedures | 2 weeks
  Dynamics according to the National Institutes of Health Stroke Scale (NIHSS) that assesses a stroke patient's impairment in a range from 0 (best score) to 42 (worst score). Details available at https://www.nihstrokescale.org/ .
Change from Baseline NIH Stroke Scale in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the National Institutes of Health Stroke Scale (NIHSS) that assesses a stroke patient's impairment in a range from 0 (best score) to 42 (worst score). Details available at https://www.nihstrokescale.org/ .
Change from Baseline American Spinal Injury Association Impairment Scale after the rehabilitation procedures | 2 weeks
  Dynamics according to the American Spinal Injury Association Impairment Scale. The scale has five classification levels from Grade A (The impairment is complete) to Grade E (The patient's functions are normal). Details available at https://asia-spinalinjury.org/international-standards-neurological-classification-sci-isncsci-worksheet/
Change from Baseline American Spinal Injury Association Impairment Scale in four weeks after the rehabilitation procedures | up to 6 weeks
  Dynamics according to the American Spinal Injury Association Impairment Scale. The scale has five classification levels from Grade A (The impairment is complete) to Grade E (The patient's functions are normal). Details available at https://asia-spinalinjury.org/international-standards-neurological-classification-sci-isncsci-worksheet/
Change from Baseline 36-Item Short Form Survey after the rehabilitation procedures | 2 weeks
  The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
  Details available at https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form.html
Change from Baseline 36-Item Short Form Survey in four weeks after the rehabilitation procedures | up to 6 weeks
  The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
  Details available at https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form.html

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Lebedev, PhD, Principal Investigator — Skolkovo Institute of Science and Technology (CNBR)
Locations (6):
- Russia (6):
  - Far Eastern Federal University, Vladivostok, Primorsky Kray
  - Samara Regional Clinical Hospital, Samara, Samara Oblast
  - Samara State Medical University, Samara, Samara Oblast
  - Kazansky Federal University, Kazan', Tatarstan Republic
  - EirMED Rehabilitation Center, Saint Petersburg
  - Pavlov Institute of Physiology, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No
Only selected research team members will have access to individual participant data. The research team will not be sharing or releasing any IPD to third parties.

REFERENCES:
- [Background] Moshonkina TR, Shapkova EY, Sukhotina IA, Emeljannikov DV, Gerasimenko YP. Effect of Combination of Non-Invasive Spinal Cord Electrical Stimulation and Serotonin Receptor Activation in Patients with Chronic Spinal Cord Lesion. Bull Exp Biol Med. 2016 Oct;161(6):749-754. doi: 10.1007/s10517-016-3501-4. Epub 2016 Oct 26. PMID 27785645
- [Background] Hofstoetter US, Hofer C, Kern H, Danner SM, Mayr W, Dimitrijevic MR, Minassian K. Effects of transcutaneous spinal cord stimulation on voluntary locomotor activity in an incomplete spinal cord injured individual. Biomed Tech (Berl). 2013 Aug;58 Suppl 1:/j/bmte.2013.58.issue-s1-A/bmt-2013-4014/bmt-2013-4014.xml. doi: 10.1515/bmt-2013-4014. Epub 2013 Sep 7. No abstract available. PMID 24042607
- [Background] Sayenko DG, Rath M, Ferguson AR, Burdick JW, Havton LA, Edgerton VR, Gerasimenko YP. Self-Assisted Standing Enabled by Non-Invasive Spinal Stimulation after Spinal Cord Injury. J Neurotrauma. 2019 May 1;36(9):1435-1450. doi: 10.1089/neu.2018.5956. Epub 2018 Dec 15. PMID 30362876
- [Background] Pichiorri F, Morone G, Petti M, Toppi J, Pisotta I, Molinari M, Paolucci S, Inghilleri M, Astolfi L, Cincotti F, Mattia D. Brain-computer interface boosts motor imagery practice during stroke recovery. Ann Neurol. 2015 May;77(5):851-65. doi: 10.1002/ana.24390. Epub 2015 Mar 27. PMID 25712802
- [Background] Lyukmanov RK, Aziatskaya GA, Mokienko OA, Varako NA, Kovyazina MS, Suponeva NA, Chernikova LA, Frolov AA, Piradov MA. [Post-stroke rehabilitation training with a brain-computer interface: a clinical and neuropsychological study]. Zh Nevrol Psikhiatr Im S S Korsakova. 2018;118(8):43-51. doi: 10.17116/jnevro201811808143. Russian. PMID 30251977
- [Background] Carvalho R, Dias N, Cerqueira JJ. Brain-machine interface of upper limb recovery in stroke patients rehabilitation: A systematic review. Physiother Res Int. 2019 Apr;24(2):e1764. doi: 10.1002/pri.1764. Epub 2019 Jan 4. PMID 30609208

DOCUMENTS (1):
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT05115149/ICF_000.pdf